CLINICAL TRIAL: NCT07346287
Title: Assessment of Symptom-Specific Improvement in Diagnosed Vaginal Atrophy Following Laser Therapy (ASSIST-VLA)
Brief Title: ASSIST-VLA: Assessment of Symptom-Specific Improvement in Diagnosed Vaginal Atrophy Following Laser Therapy
Acronym: ASSIST-VLA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Stratpharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SPAMG08
Record Dates: First submitted 2026-01-07; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Vaginal Atrophy; Atrophic Vaginitis; Genitourinary Syndrome of Menopause (GSM)
MeSH Terms: conditions — Atrophic Vaginitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Safety (Experimental)
  Interventions: Device: 7-940

INTERVENTIONS:
Device: 7-940 — A non-hormonal and non-steroidal gel that supports vulvovaginal mucosal conditions and speeds up recovery post vaginal rejuvenation. It is a suitable alternative to vaginally administered estrogen and topical corticosteroids, that promotes a moist healing environment leading to faster re-epithelialization. The gel relieves symptoms such as itchiness, tenderness, dryness, burning sensation, painful intercourse (dyspareunia), painful urination (dysuria), rectal and defecating pain. It improves erythema, mucosal tissue thinning, erosions, fissures, ulcerations, scarring/adhesions and swelling. It is indicated for long-term use to maintain the health of the vaginal mucosa without the side effects of vaginally administered hormonal therapy and topical corticosteroids.

SUMMARY:
Vaginal atrophy patients receiving vaginal laser therapy will be treated with daily 7-0940® following a laser session to evaluate the safety and efficacy of the product as an adjunct treatment. Clinical outcomes will be assessed using validated investigator- and patient-reported measures, with safety and symptom progression monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed vaginal atrophy
* Access to smartphone and tablet, laptop or computer
* Access to a valid email address
* Previously completed laser therapy session schedule

Exclusion Criteria:

* Unable to provide informed consent
* Patient unable to apply topical device
* Allergy or intolerance to ingredients or excipients of the formulation of studied products
* Systemic hormonal or steroidal therapy started less than 30 days before baseline ( = not yet on a stable regimen)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Vaginal Health Index Score (VHIS) | 30 - 45 days
  Objective clinical assessment for assessment of the device safety as adjunctive treatment after laser therapy forr women with vaginal atrophy.
  The objective validation of clinical signs (elasticity, fluid volume, pH, epithelial integrity, moisture) using a commonly used scale.
Vulvar Disease Quality of Life Index questionnaire | 30 - 45 days
  The patient-rated quality of life will be assessed at baseline and during each monthly follow-up using the validated patient-rated Vulvar Disease Quality of Life Index (VQLI). [min:0; max:45]. A higher score thereby correlates to a worse outcome. The secondary endpoint is the change from baseline VQLI score at 30 - 45 days.
Investigator-reported improvement in vaginal atrophy signs | 30-45 days
  Signs (dryness, tissue thinning, erosion, fissures, erythema, scarring, contact bleeding, labial fusion, labia reabsorption and contracture of posterior introitus) are rated by the investigator during a physical assessment at baseline and after 30 - 45 days, using a 10-point Likert scale ranging from 0=normal to 10=worst possible.
Recovery Improvement Question | 30-45 days
  Descriptive patient-related questions, assessing the improvement post-laser therapy.

SECONDARY OUTCOMES:
Change in complication rate | 30 - 45 days
  Any adverse reactions or complications, are rated by the investigator during each assessment baseline and after 30 - 45 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Orange Coast Women's Medical Group, Laguna Hills, California, United States